CLINICAL TRIAL: NCT01308502
Title: A New Nasopharyngeal pH Probe for Diagnosis of Laryngopharyngeal Reflux
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting patients due to logistics
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Karen Zur, Associate Director, The Center for Pediatric Airway Disorders, Director Pediatric Voice Program, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-007341
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Laryngopharyngeal Reflux
Keywords: laryngopharyngeal reflux; LPR; GERD; gastroesophageal reflux; nasopharyngeal probe
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probe (Experimental): Children with airway obstruction
  Interventions: Device: Dx-pH probe

INTERVENTIONS:
Device: Dx-pH probe — Dx-pH probe with 24 hour recording
  Other Names: ResTech Dx-pH probe

SUMMARY:
The purpose of this study is to evaluate the utility of a minimally invasive nasopharyngeal pH probe for the diagnosis of laryngopharyngeal reflux (LPR) in children with airway compromise; to determine whether it is comparable to the gold standard esophageal pH probe in identifying LPR in this population; and to correlate results of pH testing with validated questionnaires. Our hypothesis is that a nasopharyngeal pH probe is equivalent to an esophageal probe in identifying laryngopharyngeal reflux.

DETAILED DESCRIPTION:
Laryngopharyngeal reflux (LPR) has been repeatedly linked to upper respiratory symptoms in the pediatric population. Children with LPR may present with laryngomalacia, subglottic stenosis, laryngitis, and vocal cord nodules among other illnesses. Pharyngeal reflux has even been implicated in causing common childhood illnesses such as sinusitis and otitis media. Diagnosing LPR can be difficult, especially in children. Often otolaryngologists depend on a general gestalt to diagnosis LPR. In some cases, physicians rely on a Reflux Symptoms Index (RSI) questionnaire filled out by the caretaker and/or a Reflux Finding Score (RFS) filled out by the practitioner. Others have attempted to use a variety of tools to measure pH in the upper airway and proximal esophagus.

Initial research focused on correlating gastroesophageal reflux (GER) with otolaryngologic illnesses. These studies relied mostly on esophageal pH probes placed at the lower esophageal sphincter. With the realization that extraesophageal reflux or LPR was a separate disease, new methods have developed to quantify it. The dual esophageal pH probe is the current gold standard for measuring LPR as it records pH just above the proximal esophageal sphincter. Conditions such as chronic pediatric sinusitis, otitis media, laryngitis and globus are believed to arise from laryngopharyngeal reflux. Unfortunately, this device fails to identify many patients with LPR who would benefit from treatment, and radiographic studies are limited by their short duration of evaluation and risk of radiation. In addition, the placement of the esophageal pH probe is relatively invasive requiring both sedation and x-rays to confirm placement. Finally, they are difficult to place and maintain in children, necessitating a hospital stay for 24 hours while data is collected. The alternative is empiric treatment with Histamine 2 blockers and/or Protein Pump Inhibitors for an extended course, which has been shown to improve symptoms in many of these patients but is not without risk.

The new Dx-pH nasopharyngeal probe is the only tool available for directly measuring nasopharyngeal pH. It is an exempted class I medical device and is Food and Drug Administration (FDA)-approved for general use in the population. The device, manufactured by Respiratory Technology Corporation ISO (ResTech), measures the pH of both liquid and aerosolized droplets. It is positioned posterior to the soft palate and placement is confirmed by visualizing the light-emitting diode (LED) at the tip of the device. It is significantly less invasive than esophageal pH probes, does not require general anesthesia for placement, and can be used in an outpatient setting.

The Dx-pH probe is currently being used clinically in adult and pediatric practices to diagnose and monitor laryngopharyngeal reflux with only limited research supporting its use. A literature review finds only 6 studies that address the Dx-pH probe, of which, only 1 pilot study has been performed in children. This study looked at changes in pH in the trachea of 3 children with chronic tracheostomies. However, to date, no research has been published on the utility of the probe in diagnosing LPR in children. The probe, if effective, would be a valuable tool for diagnosing LPR in the pediatric population because of its limited risk and potential ability to replace more invasive and costly procedures.

ELIGIBILITY:
Inclusion Criteria:

* History of airway compromise
* Undergoing microlaryngoscopy, bronchoscopy, esophagoscopy, and esophageal pH probe placement at CHOP

Exclusion Criteria:

* Patients not undergoing esophageal pH probe placement
* Neonates under 1 month of age
* Adults over 18 years of age or older.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
nasopharyngeal pH | 24 hours
  Change in nasopharyngeal pH as measured by the Dx-pH probe

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zur, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States